CLINICAL TRIAL: NCT01742520
Title: Its an Interventional Study That Will Evaluate the Effect of Different Doses of Sucrose 24% on Neurodevelopmental Outcome of Preterm Infants
Brief Title: Neurodevelopmental Outcomes of Preterm Infants Treated for Pain Management With Repeated Doses of Sucrose 24%
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Iris Morag, Staff Neonatologist, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-12-9389-IM-CTIL
Record Dates: First submitted 2012-11-18; First posted 2012-12-05 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Development
Keywords: Preterm infant; pain; neurodevelopment
MeSH Terms: conditions — Premature Birth; Pain | interventions — Food, Formulated; Milk, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formula or Breast Milk (Active Comparator): Breast milk or formula prior to every painful procedure.
  Interventions: Drug: Formula or breast milk
- Multiple doses of sucrose (Active Comparator): Infants in this group will be treated with Sucrose 24% 0.5-1ml on the anterior pat of the tongue 1-3min prior to every invasive procedure
  Interventions: Drug: multiple doses of sucrose

INTERVENTIONS:
Drug: multiple doses of sucrose — unlimited number of doses par day- current status in our NICU
  Other Names: sucrose 24%
  Arms: Multiple doses of sucrose
Drug: Formula or breast milk — 1-3 minutes prior to every painful procedure, breast milk or formula 0.5-1 ml will be given on the anterior part of the tongue
  Other Names: sucrose 24%
  Arms: Formula or Breast Milk

SUMMARY:
The purpose of this study is to determine the effect of sucrose 24% for pain prevention on preterm infants. Our hypothesis is that repeated doses of sucrose 24%, given prior to painful procedure,do not impair neurodevelopmental outcomes of preterm infants

DETAILED DESCRIPTION:
preterm infants born at 27-33 weeks gestational age at Sheba Medical Center will be recruited for this study. Prior to invasive procedure infants will be treated with pacifier and swaddling as recommended by the American Academy of Pediatrics and Canadian Pediatric Society.

Group 1.Will be treated with Sucrose 24% 0.1-0.5ml on the anterior pat of the tongue 1-3 min prior to invasive procedure.

Group 2. Similar to group 1 but breast milk or formula will replace Sucrose.

Number of invasive procedures/day will be documented

General Movements by Prechtel will be used for developmental assessment at 2,4,6 weeks after birth and at 14-16 weeks corrected age

Griffiths developmental scales (GMDS) will be used at 40 weeks, 14-16 weeks corrected age, and 3-6 month corrected age

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born at SMC

Exclusion Criteria:

* need for intubation
* surgery
* need for sedation
* abnormal head ultrasound
* genetic abnormalities
* necrotizing enterocolitis
* other painful conditions other than routine blood exams

Ages: 27 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
neurodevelopmental outcomes | at 6 month corrected age
  Griffith mental developmental scaled (gross and fine motor, language, performance, social) and General movements by Prechtel

SECONDARY OUTCOMES:
neurodevelopment | at 15 weeks corrected age
  Griffith mental developmental scaled (gross and fine motor, language, performance, social) and General movements by Prechtel

CONTACTS AND LOCATIONS:
Overall Officials: Iris Morag, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Result] Johnston CC, Filion F, Snider L, Majnemer A, Limperopoulos C, Walker CD, Veilleux A, Pelausa E, Cake H, Stone S, Sherrard A, Boyer K. Routine sucrose analgesia during the first week of life in neonates younger than 31 weeks' postconceptional age. Pediatrics. 2002 Sep;110(3):523-8. doi: 10.1542/peds.110.3.523. PMID 12205254